CLINICAL TRIAL: NCT00030667
Title: A Phase II Study of Gleevec (Imatinib Mesylate, NSC 716051 Formerly STI571) in Children With Refractory or Relapsed Solid Tumors
Brief Title: Imatinib Mesylate in Treating Patients With Relapsed or Refractory Solid Tumors of Childhood
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01869; NCI-2012-01869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069187; COG-ADVL0122; ADVL0122 (Other: Children's Oncology Group); ADVL0122 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2002-02-14; First posted 2003-05-07 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2013-12

CONDITIONS: Childhood Desmoplastic Small Round Cell Tumor; Childhood Synovial Sarcoma; Gastrointestinal Stromal Tumor; Lung Metastases; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Neuroblastoma; Recurrent Osteosarcoma
MeSH Terms: conditions — Desmoplastic Small Round Cell Tumor; Gastrointestinal Stromal Tumors; Neuroectodermal Tumors, Primitive, Peripheral; Neuroblastoma; Osteosarcoma | interventions — Imatinib Mesylate

ARMS (1):
- Treatment (imatinib mesylate) (Experimental): Patients receive oral imatinib mesylate once or twice daily on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: imatinib mesylate; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of imatinib mesylate in treating patients who have relapsed or refractory solid tumors of childhood. Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate of patients with relapsed or refractory pediatric solid tumors treated with imatinib mesylate.

II. Determine the toxicity of this drug in these patients. III. Determine the time to progression in patients treated with this drug. IV. Determine the pharmacokinetics of this drug in these patients. V. Correlate response with c-kit and platelet-derived growth factor receptor expression in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (Ewing's sarcoma/primitive neuroectodermal tumor vs osteosarcoma vs neuroblastoma vs other).

Patients receive oral imatinib mesylate once or twice daily on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumors including the following:

  * Ewing's sarcoma
  * Bone or soft tissue primitive neuroectodermal tumor
  * Osteosarcoma
  * Neuroblastoma
  * Desmoplastic small round cell tumor
  * Synovial cell sarcoma
  * Gastrointestinal stromal tumor (GIST)
* Metastatic pulmonary disease eligible

  * No pleural effusion of any size or definite radiologic evidence of pleural-based disease
* Recurrent or refractory to conventional therapy

  * GIST eligible at initial presentation
* Tumor tissue blocks must be available
* At least 1 measurable lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * Lesions assessable only by radionuclide scan are not considered measurable
* Performance status - Lansky 50-100% (≤ 10 years of age)
* Performance status - Karnofsky 50-100% (> 10 years of age)
* At least 2 months
* Absolute neutrophil count ≥ 1,000/mm^3*
* Platelet count ≥ 75,000/mm^3* (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL* (RBC transfusions allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN
* INR < 1.5
* PTT ≤ ULN
* Fibrinogen ≥ lower limit of normal
* Creatinine normal for age
* Glomerular filtration rate ≥ 70 mL/min
* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* At least 1 week since prior biologic therapy or immunotherapy and recovered
* At least 1 week since prior growth factors
* No concurrent immunomodulating agents
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No concurrent chemotherapy
* No concurrent steroids
* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 3 months since prior craniospinal radiotherapy or radiotherapy to 50% or more of pelvis
* At least 6 weeks since other prior substantial bone marrow radiation
* No concurrent radiotherapy during first course of treatment
* Concurrent palliative radiotherapy to local painful lesions allowed after first course of treatment provided there is no evidence of disease progression and at least 1 measurable lesion remains outside radiation port
* No concurrent therapeutic doses of warfarin
* No concurrent anticonvulsants that induce the cytochrome p450 enzyme system (e.g., phenytoin, carbamazepine, and phenobarbital)
* Concurrent benzodiazepines and gabapentin allowed
* Concurrent low-molecular weight heparin allowed

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2002-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Response rate, determined using the RECIST criteria | Up to 2 years
  95% confidence interval will be computed.
Toxicity reported using the CTC version 2.0 | Up to 2 years

SECONDARY OUTCOMES:
Time to disease progression | Up to 2 years
  Calculated by the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Mason Bond, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States